CLINICAL TRIAL: NCT06323954
Title: Pairing tVNS With Motor Skill Training in Older Adults
Brief Title: tVNS During Motor Training in Older Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Georgia Institute of Technology (Other)
Collaborators: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: H24110
Record Dates: First submitted 2024-03-15; First posted 2024-03-21 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-03

CONDITIONS: Older Adults

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tVNS stimulation (Experimental): Brief electrical current will be applied to the vagus nerve area (the tragus or cymba concha, depending on the shape and size of the ear) immediately after successful trials during finger control training.
  Interventions: Procedure: tVNS stimulation
- Sham stimulation (Sham Comparator): Brief electrical current will be applied to the non-vagus nerve area (the earlobe) immediately after successful trials during finger control training.
  Interventions: Procedure: Sham stimulation

INTERVENTIONS:
Procedure: tVNS stimulation — Electrical stimulation to the vagus nerve area.
  Arms: tVNS stimulation
Procedure: Sham stimulation — Electrical stimulation to the non-vagus nerve area.
  Arms: Sham stimulation

SUMMARY:
The goal of this study is to learn about the effect of applying transcutaneous vagus nerve stimulation (tVNS) during motor training on motor learning in older adults. The main question it aims to answer is whether applying tVNS after successful motor trials (post-success tVNS) will facilitate the rate of motor learning. Participants will be randomly assigned to tVNS or sham group and receive tVNS or sham, respectively, at the outer ear during finger control training sessions. Finger control performance will be tested before and after the training sessions without outer ear stimulation.

DETAILED DESCRIPTION:
The participants will be randomly assigned to a tVNS or control group. They will visit the lab for four sessions. The main motor task is to trace target trajectories with finger forces. As the pre- and post-tests, all participants will be tested on a force tracing motor task with the left hand. There will be no electrical stimulation during the tests. During the training sessions, all participants will wear surface electrodes on the outer ear. The attachment sites are the tragus or cymba concha (depending on the shape and size of the ear) for the tVNS group and the earlobe for the sham group. The participants will perform finger training to trace target trajectories with their left finger forces. Participants in the tVNS and sham group will receive tVNS and sham stimulation, respectively, after successful finger trials.

ELIGIBILITY:
Inclusion Criteria:

* 65-84 years old across all races, genders, and ethnicities.
* Right-handed
* Physically and cognitively healthy

Exclusion Criteria:

* Younger than 65 years old or older than 84 years old
* Current or history of cardiac disease
* Have an implanted device such as a neurostimulator or cochlear implant
* Current or history of tympanic membrane perforation
* Have a musculoskeletal issue that prevents hand function (e.g., arthritis)
* Have a vision problem not corrected by glasses or contact lenses
* Uncorrected auditory impairments
* Had a stroke or lesion (including tumor) in the brain
* Had a head injury or brain surgery
* Suffer from frequent or severe headaches
* Had a fainting spell or syncope
* Have any metal in the head such as shrapnel, surgical clips, or fragments from welding or metal work
* Have any implanted device such as cardiac pacemakers, medical pumps, or intracardiac lines
* Had any brain-related conditions (i.e. multiple sclerosis, Parkinson, Alzheimer)
* Had any illness that caused brain injury (i.e. meningitis, aneurysm, brain tumor)
* Had any head trauma that was associated with a loss of consciousness or diagnosed as a concussion
* Being treated for any psychiatric condition (i.e. depression, anxiety, PTSD, schizophrenia)
* Suspected of pregnancy
* Pregnant
* Cognitive status issues as confirmed with the Mini-Mental State Exam (MMSE <26)
* Musculoskeletal condition or injury that would limit hand range of motion

Ages: 65 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-05-27 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Rate of error reduction | 2 weeks
  The slope of the reduction in the root mean square error of finger force

CONTACTS AND LOCATIONS:
Overall Officials: Minoru Shinohara, PhD, Principal Investigator — Georgia Institute of Technology
Locations (1):
- Human Neuromuscular Physiology Lab, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided